CLINICAL TRIAL: NCT05305807
Title: Effect of Postural Correction Exercises on Shoulder Muscles Tenderness and Performance in Subjects Addicting Smartphones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasha Magdy Ibrahim Mohamed, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003350
Record Dates: First submitted 2022-02-26; First posted 2022-03-31 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Ergonomics
Keywords: Smartphone addiction; Shoulder mechanics
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Postural exercises will be done to this group
  Interventions: Other: Postural exercises
- Control group (No Intervention): Postural exercises will not be done to this group

INTERVENTIONS:
Other: Postural exercises — Postural correction exercises are effective in improving forward head posture and it effectively decrease neck pain and increase ROM Exercise training and ergonomic guidelines concerning the use of touchscreen smartphones will reduce the risk of developing upper extremity musculoskeletal disorders
  Arms: Study group

SUMMARY:
smartphones have replaced most of the keypad phone products due to their small size and easy of portability. As a result, smartphone users experience an increase in musculoskeletal problems in the neck and shoulder. Therefore, the importance of exercise and proper training should be emphasized for people who are likely to develop postural deformities due to incorrect posture habits and daily living patterns

DETAILED DESCRIPTION:
Prolonged VDTs operation is a leading cause of musculoskeletal disorders and cumulative trauma disorders such as stiff shoulders, neck soreness, carpal tunnel syndrome, and low back pain among office employees. The problems are intensified by wrong work postures, such as flexed neck, wrists, or excessively flexed forearms.Smartphone is a mobile hand-held VDT device with advanced computing capability, such as internet communication, information retrieval, video display and other capabilities. Being portable, smartphones have had a large impact on modern everyday life on terms of inducing continuous mechanical stress on shoulder and neck tendons and muscles caused by it's prolonged use.

Attaining ideal posture puts least stress on spinal structures. A good posture of head and shoulder is attaining by keeping ears aligned with the shoulders and shoulder joints retracted. Person attaining ideal posture put least stress on spinal structures. The commonest posture adapted by smartphone users is bending their neck and staring at the mobile screen, which subsequently causes postural alteration and leads to neck pain. It is found that there is extremely significant correlation between prolonged use of smartphone and forward head posture.

Posture correction exercises correct postural alterations like forward head posture and rounded shoulder posture. It is found that deep neck flexors, isometric extension, prone chin tucks and chest stretches are effective in correcting forward head posture by improving craniovertebral angle. Scapular stabilization exercises are found to be effective in increasing shoulder range of abduction and external rotation and in decreasing forward head and shoulder postures.

ELIGIBILITY:
Inclusion Criteria:

1. Forty-two subjects of both sexes will be recruited in the study.
2. The age range of the recruited subjects will be ranging from 25 to 34 years old.
3. For objective assessment of smartphone addiction, smartphone addiction scale will be made
4. Recruited subjects will be selected based on having postural deviation in the form of rounded shoulders (CVA is less than 45°) (Weon et al.,2010) and forward head posture( shoulder angle more than 35°

Exclusion Criteria:

1 - Subjects with history of previous injury of the neck, shoulder. 2-Subjects with history of surgical intervention at the neck or upper extremity.

3-Subjects with history of inflammatory joint disease affecting shoulder and facet joints.

4-Subjects with musculoskeletal disorders related to neck or upper limb such as rotator cuff tendinitis and impingement syndrome.

5-Subjects with neurological disorders that affect upper limb muscular performance such as cervical spondylosis, spondylolythesis, disc prolapse or thoracic outlet syndrome.

6-Athletes who practice sports that require use of shoulder muscular group such as volleyball, basketball, boxing.

Ages: 25 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Shoulder muscles peak torque | 4 weeks
  Newton.meter
Shoulder muscles work | 4 weeks
  Joules
Shoulder muscles work fatigue | 4 weeks
  Joules
Shoulder muscles pain threshold | 4 weeks
  Newton

CONTACTS AND LOCATIONS:
Overall Officials: Ragia MO Kamel, Ph.D, Study Chair — Professor of Physical Therapy-Cairo university; Amr SA Shalaby, Ph.D, Study Director — Professor of Physical Therapy-Cairo University
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol
Time Frame: Within six months of termination of the current study
Access Criteria: IPD sharing will be done after publication of the study results.